CLINICAL TRIAL: NCT03863132
Title: Optimal Medical Treatment With or Without Valve Repair in Patients With Symptomatic Paradoxical Low-Flow, Low-Gradient Aortic Stenosis - a Multi-center, Randomized Comparison
Brief Title: accuRate Evaluation of Benefit With Optimal Medical Treatment With or Without Transcatheter Valve Repair of PARADOXical Low Flow Low Gradient Aortic Stenosis
Acronym: REBOOT-PARADOX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Collaborators: Boston Scientific Group (Unknown); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REBOOT-PARADOX
Record Dates: First submitted 2019-02-27; First posted 2019-03-05 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic stenosis; Low flow; Low gradient; Transcatheter aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, randomized (2:1), parallel group, open-label, multi-centre, international
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAVR Group (Active Comparator): Patients will be treated by transcatheter aortic valve repair (TAVR).
  Interventions: Device: TAVR
- Medical Treatment Group (No Intervention): Patients will receive optimal medical treatment alone.

INTERVENTIONS:
Device: TAVR — Repair of defective aortic valve by microsurgical Intervention.
  Arms: TAVR Group

SUMMARY:
Aim of this study is to evaluate whether microsurgical repair or replacement of the aortic valve is a treatment option for a subgroup of patients suffering from aortic Stenosis.

DETAILED DESCRIPTION:
Stenosis of the aortic valve leads to a narrowing of the valve, consequently to low blood flow from the heart into the Aorta, and is associated with symptoms like fatigue, breathlessness, dizziness, fainting, and chest pain. For many of the patients suffering from severe aortic stenosis surgical or catheter-assisted repair or replacement of the damaged aortic valve has been proven to be a safe and effective treatment option.

Probably about 20-30% of patients suffering from severe aortic stenosis display a deviation from the usually observed disease pattern: These patients do not show the typical high pressure difference between the left ventricle (heart chamber) and the aorta (transvalvular gradient; "paradoxical" low flow/low gradient aortic stenosis). For these patients it is not yet clear, if microsurgical repair of the aortic valve (transcatheter aortic valve repair - TAVR) should be a treatment option as well.

REBOOT-PARADOX evaluates whether TAVR is advantageous compared to optimal medical Treatment alone for patients suffering from paradoxical aortic stenosis. Two thirds of the participating patients will be treated by TAVR, one third will receive medical Treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* I1. Patients with symptomatic native aortic valve stenosis and age ≥18 years
* I2. Aortic valve area (AVA) ≤ 1 cm2 or indexed AVA ≤ 0.6 cm2/m2, mean aortic gradient < 40 mmHg and stroke volume index (SVI) < 35ml/m2
* I3. Left ventricular ejection fraction ≥ 50%
* I4. MDCT aortic valve calcium score men > 2000AU, women > 1200AU OR the likelihood criteria are fulfilled (symptoms without other explanation and LV hypertrophy; age < 70 yrs., AVS < 0.8 cm2; SVI < 35ml/m2 confirmed by 3D TOE, MRI or invasive; reduced LV longitudinal function without other reason)
* I5. Heart team agrees on eligibility for TAVR
* I6. Written informed consent
* I7. Negative pregnancy test in women with childbearing potential

Exclusion Criteria:

* E1. Hemodynamic instability
* E2. Cardiogenic shock
* E3. Pre-existing mechanical or bio-prosthetic valve in any position
* E4. Concomitant severe valvular heart disease
* E5. Pre-existing or active endocarditis
* E6. Need for heart surgery due to other conditions
* E7. Aortic valve is congenital unicuspid or congenital bicuspid
* E8. Hypertrophic cardiomyopathy with or without obstruction
* E9. Echocardiographic evidence of intracardiac mass, thrombus or vegetation
* E10. Acute myocardial infarction within 1 month before intended AS-treatment
* E11. Renal replacement therapy
* E12. Estimated life expectancy < 24 months (730 days) due to carcinomas end stage liver disease or renal disease
* E13. Currently participating in an investigational drug or another device study. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
* E14. Patient refuses aortic valve repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Time to death | 24 months after last-patient-in
  All-cause mortality

SECONDARY OUTCOMES:
Cardiovascular mortality | 5 years after index treatment
  Death because of cardiovascular events
Re-hospitalization due to heart failure | 5 years after index treatment
  Number of hospital stays after randomization
Incidence of neurological events - incidence of strokes | 5 years after randomization
  Number of strokes
Incidence of neurological Events - incidence of transient ischaemic attacks | 5 years after randomization
  Number of transient ischaemic attacks
Cardiac functionality - left ventricular function | 5 years after randomization
  Echocardiographic measurement of left ventricular ejection fraction in %
Cardiac functionality - aortic valve hemodynamics | 5 years after randomization
  Measurement of aortic pressure in mmHg
Patients' quality of life | 5 years after randomization
  EQ5D-score in %
Device reliability | 5 years after randomization
  Number of reinterventions (TAVR arm only)

CONTACTS AND LOCATIONS:
Overall Officials: Julinda Mehilli, Prof. Dr., Principal Investigator — University Clinic Munich
Locations (1):
- Klinikum der Universität München-Großhadern, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No